CLINICAL TRIAL: NCT04436835
Title: Accelerated Resolution Therapy for Cancer Related Trauma and Distress: a Pilot Study
Brief Title: Psychotherapy (Accelerated Resolution Therapy) for Cancer Related Trauma and Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cindy Tofthagen, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-006093; NCI-2020-04130 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-006093 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (ART) (Experimental): Patients undergo ART over 60-90 minutes once a week for up to 5 sessions.
  Interventions: Behavioral: Psychotherapy; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Psychotherapy — Undergo ART
  Other Names: talk therapy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies whether a form of psychotherapy called accelerated resolution therapy can help with cancer distress and psychological trauma. Accelerated resolution therapy is an evidence-based therapy for the treatment of depressive symptoms, trauma, and stress-related disorders. This study may provide evidence to support integration of accelerated resolution therapy into psychological treatment of cancer patients, which may decrease cancer related trauma and distress.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Calculate changes, and estimate mean changes, in primary outcomes of psychological trauma and cancer distress over a six week time period while receiving weekly accelerated resolution therapy (ART).

II. Calculate changes, and estimate mean changes, in secondary outcomes of anxiety and depression over a six week period while receiving weekly ART.

III. Will use a qualitative, descriptive design to explore contextual elements of the cancer experience that are consistently distressing and/or psychologically traumatic to more fully inform a future RCT testing in ART in cancer distress and psychological trauma.

IV. Calculate changes, and estimate mean changes, in secondary outcomes of resilience and symptom distress over a six week period while receiving weekly ART.

OUTLINE:

Patients undergo ART over 60-90 minutes once a week for up to 5 sessions.

After completion of study intervention, patients are followed up at 1 week and again at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write and understand English
* Undergone chemotherapy, radiation therapy, chimeric antigen receptor T cells (CAR-T), or bone marrow transplant for a cancer diagnosis within the previous 3 years or have metastatic cancer
* A mean score of at least 1.1 on the Cancer and Treatment Distress (CTxD) or at least one item rated at a 3 (often true) or 4 (nearly all the time)
* A minimum score of 3 on the Primary Care-Post Traumatic Stress Disorder Screen (PC-PTSD-5)
* Denial of suicidal ideation or intent, with no evidence of psychotic behavior
* Participants must be willing and able to utilize secure web conferencing software, phone calls, or to travel to Mayo Clinic outside of normally scheduled visits to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Psychological trauma | Up to 6 weeks
  Symptoms of psychological trauma will be measured with both the Primary Care-Post Traumatic Stress Disorder Screening (PC-PTSD-5) and the Post Traumatic Stress Disorder Checklist (PCL-5). The PCL-5 (PTSD Patient Checklist) is a 20-item self-report instrument that will be used to assess the DSM-5 symptoms of PTSD (psychological trauma). The total symptom severity score ranges from 0 to 80.
Cancer distress | Up to 6 weeks
  Cancer distress will be measured with the Cancer Treatment Distress Scale (CTxD). The CTxD is a 22 item Likert type scale that contains 6 subscales: uncertainty, health burden, identity, medical demands, finances, and family strain. Scores on individual items range from 0 (none) to 3 (severe) distress related to an aspect of the cancer experience.

SECONDARY OUTCOMES:
Anxiety | Up to 6 weeks
  The General Anxiety Disorder (GAD-7) is a measure of anxiety scored from 0 (not at all)-3 (nearly every day) scale for each item with total scores ranging from 0-21. A score of 10 or more indicates high anxiety, although a cut-score of 7 or higher has been suggested for cancer populations.
Depression | Up to 6 weeks
  The Patient Health Questionnaire (PHQ-8) is an 8 item measure of depression scoring DSM -IV criteria for depression on a 0 (not at all) to 3 (nearly every day) scale for each item with total scores ranging from 0-24 (25). A score of 10 or more indicates depression.
Resilience | Up to 6 weeks
  The Connor-Davidson Resilience Scale (CD-RISC) is a 10 item scale in which participants rate statements on a scale of 0 (not at all true) to 4 (true nearly all the time). Higher scores indicate higher levels of resilience.
Symptom distress | Up to 6 weeks
  The Edmonton Symptom Assessment Scale (ESAS) consists of 11-point numerical rating scales for self-report of ten common symptoms of cancer. A summary score is calculated with higher scores representing greater symptom distress.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Tofthagen, Ph.D., R.N., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials